CLINICAL TRIAL: NCT04709003
Title: Covid-19 Vaccine Effectiveness in Healthcare Personnel in Clalit Health Services in Israel (CoVEHPI): A Prospective Cohort Study
Brief Title: Covid-19 Vaccine Effectiveness in Healthcare Personnel in Clalit Health Services in Israel (CoVEHPI)
Acronym: CoVEHPI
Status: Completed | Type: Observational
Sponsor: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Ran Balicer, Chief Innovation Officer, Clalit Health Services, Clalit Health Services
Other Study IDs: 1051-20-RMC-C
Record Dates: First submitted 2021-01-06; First posted 2021-01-14 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Covid19; Corona Virus Infection; Vaccine Effectiveness
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Serologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vaccinated: participants who received the Covid-19 vaccine
  Interventions: Diagnostic Test: Serologic test; Diagnostic Test: Respiratory swabs
- unvaccinated: participants who didn't received the Covid-19 vaccine
  Interventions: Diagnostic Test: Serologic test; Diagnostic Test: Respiratory swabs

INTERVENTIONS:
Diagnostic Test: Serologic test — A blood test to check antibodies type and amount
Diagnostic Test: Respiratory swabs — PCR test to Covid-19

SUMMARY:
Although clinical trials for approved COVID-19 vaccines demonstrated efficacy of the vaccine in preventing symptomatic infection, many questions about vaccine effectiveness, such as the effectiveness of COVID-19 vaccine in preventing asymptomatic infection, a surrogate for transmission, and duration of protection, can only be evaluated in real-world trials. The objective of the study is to evaluate COVID-19 vaccine effectiveness (Pfizer vaccine, and, if available, Moderna vaccine) in preventing infection in healthcare personnel in Israel. HCP who are Clalit members and working in Soroka, Beilinson, Meir, Haemek, Kaplan and Schneider hospitals, 18 years or older, and eligible to get COVID-19 vaccine according to Ministry of Health guidelines, will be recruited, regardless of their intention to get the COVID-19 vaccine. A baseline serology sample and respiratory sample will be collected. Participants will be asked to provide a respiratory sample weekly for 3 months, and then monthly for the remainder of the study. Participants will also have blood drawn at 1 month, 3 months, 6 months, 9 months and 12 months. Respiratory samples will be tested for SARS-CoV-2 by RT-PCR; serology will be tested for SARS-CoV-2 antibodies. The study will last for 12 months. For each participant, data will be extracted from the Electronic Medical Record for the period of the study and retrospectively from 2010.

ELIGIBILITY:
Inclusion Criteria:

- Any HCP at any of the participating hospitals who is

* a member of Clalit Health Services
* is eligible to get the Covid-19 vaccine
* did not receive the first dose of COVID-19 vaccine more than 21 days prior to the enrollment date

Exclusion Criteria:

-

Employees at any of the participating hospitals will be excluded if they are:

* not a member of Clalit Health Services; or
* not eligible to get the Covid-19 vaccine according to the Ministry of Health guidelines; or
* Less than 18 years of age
* Received first dose of COVID-19 vaccine more than 21 days prior to date of enrollment

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare workers who work in 6 Clalit hospitals in Israel (Soroka, Kaplan, Meir, Beilinson, HaEmek, and Schneider)
Sampling Method: Non-Probability Sample
Enrollment: 1567 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
COVID-19 vaccine effectiveness (VE) | 18 months
  Incidence of SARS-CoV-2 infections in healthcare workers vaccinated with COVID-19 vaccine compared to unvaccinated healthcare workers

SECONDARY OUTCOMES:
Symptomatic SARS-CoV-2 infection in vaccinated vs. unvaccinated healthcare workers | 18 months
  Incidence of symptomatic SARS-CoV-2 infections in healthcare workers vaccinated with COVID-19 vaccine compared to unvaccinated healthcare workers
asymptomatic SARS-CoV-2 infection in vaccinated vs. unvaccinated healthcare workers | 18 months
  Incidence of symptomatic SARS-CoV-2 infections in healthcare workers vaccinated with COVID-19 vaccine compared to unvaccinated healthcare workers
Duration of effectiveness of the vaccine | 18 months
  Incidence of SARS-CoV-2 infections in healthcare workers vaccinated with COVID-19 vaccine compared to unvaccinated healthcare workers over different periods of time
Vaccine Effectiveness by age | 18 months
  Incidence of SARS-CoV-2 infections in healthcare workers vaccinated with COVID-19 vaccine compared to unvaccinated healthcare workers of different age groups
Vaccine Effectiveness by comorbidity | 18 months
  Incidence of SARS-CoV-2 infections in healthcare workers vaccinated with COVID-19 vaccine compared to unvaccinated healthcare workers by various underly medical conditions
Vaccine effectiveness in persons previously infected with SARS-CoV-2 virus | 18 months
  Incidence of SARS-CoV-2 infections in previously infection healthcare workers vaccinated with COVID-19 vaccine compared to previously infection unvaccinated healthcare workers
VE by degree of exposure to COVID-19 patients | 18 months
  Incidence of SARS-CoV-2 infections in healthcare workers vaccinated with COVID-19 vaccine compared to unvaccinated healthcare workers by degree of occupational exposure to COVID-019 patients
VE by different SARS-CoV-2 variants | 18 months
  Incidence of SARS-CoV-2 infections in healthcare workers vaccinated with COVID-19 vaccine compared to unvaccinated healthcare workers for different variant strains of SARS-CoV-2
Vaccine effectiveness of one dose compared to two doses | 18 months
  Incidence of SARS-CoV-2 infections in healthcare workers vaccinated with two doses of COVID-19 vaccine compared to healthcare workers vaccinated with two doses of COVID-19 vaccine
Compartive vaccine Effectiveness of different vaccine brands | 18 months
  Incidence of SARS-CoV-2 infections in healthcare workers vaccinated with different brands of COVID-19 vaccine

CONTACTS AND LOCATIONS:
Locations (6):
- Israel (6):
  - Haemek Medical Center, Afula
  - Soroka Medical Center, Beersheba
  - Meir Medical Center, Kfar Saba
  - Beilinson hospital, Petah Tikva
  - Schneider Children's Medical Center of Israel, Petah Tikva
  - Kaplan Medical Center, Rehovot

IPD SHARING:
Plan to Share IPD: Undecided